CLINICAL TRIAL: NCT00462683
Title: Bone Loss, Fractures, and Management of Bone Health in People With Stroke in Managed Rehabilitation Settings
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, professor, Northwestern University
Other Study IDs: NURIC0445100
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Stroke; Anoxia; Brain Injury
Keywords: Stroke; Anoxia; Brain Injury; Rehabilitation; Osteoporosis; Osteopenia
MeSH Terms: conditions — Stroke; Hypoxia; Brain Injuries; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two 10ml tubes of blood will be obtained from each participant. Serum will be separated and frozen to be saved for possible measurement of vitamin D levels and/or bone markers.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate the state of bone health of brain injury patients being seen within a rehabilitation setting. Osteopenia is a condition of bone in which decreased calcification, decreased density, or reduced mass occurs. Osteoporosis is a disease in which the bones become extremely porous, are subject to fracture, and heal slowly. More specifically, the prevalence of osteopenia and osteoporosis at specific anatomic locations (e.g., forearms, hips, spine) will be determined as will specific interventions (e.g., use of vitamins, nutritional supplements, specific prescription medications) that people with brain injury may be applying, or have applied, to manage their bone health. An attempt will also be made to evaluate severity of brain injury, based on loss of muscle strength/function, and to compare this data with bone-focused information such as bone mineral density (BMD), falls, and history.

DETAILED DESCRIPTION:
Primary Outcomes: As this study has no control or comparator group, the goal will be to provide descriptive data regarding the prevalence of osteopenia and osteoporosis at each of the anatomic sites evaluated by DEXA in this specialized population (BMD outcome measures). Additionally, the use of bone-specific interventions (vitamins, nutritional supplements, medications), previous diagnostic testing (DEXA) and history of falls and fractures will be assessed to determine the extent to which bone health has been considered and evaluated in this population of individuals at increased risk of fracture.

Secondary Outcomes: Functional status measures will also be obtained to enable correlation with bone data.

This study involves a cross-sectional, descriptive evaluation of a cohort of 225 patients with brain injury who are being managed at the out-patient clinics by physicians from RIC. The goal of the study is to provide representative data of both the general bone health of this population of patients (degree, extent and localization of bone loss) as well as interventions that may have been implemented to manage their bone health (vitamins, nutritional supplements, prescription medications). After obtaining informed consent, those patients who wish to be involved will be asked to complete a medical history questionnaire that focuses on bone health and will then undergo measurement of bone density by DEXA (dual energy X-ray absorptiometry). At the time of the DEXA examination, muscle strength will be evaluated by a trained research coordinator. A dietary history and a blood sample will also be obtained, the latter for storage in order to later measure vitamin D levels and/or other bone markers. All subjects will then be given the opportunity to continue in the longitudinal arm of the study (second phase). Those who do will sign the informed consent and will then be re-evaluated at yearly intervals with the same set of data being obtained.

Descriptive Data to be Obtained:

1. Demographics: date of birth, sex, race, ethnicity
2. Detailed and complete medical history, with particular focus on:

   * Information regarding brain injury: time of occurrence, motor/sensory, etc.
   * Bone specific information: history of falls, fractures, use of medications, smoking, alcohol, family history of osteoporosis and fractures, previous DEXA, etc.
   * Questionnaire of functional status: use of affected arm, ambulation, assistive device, orthotic, frequency of spasms.
   * Evaluation of motor status using the Motor Components of the NIH Stroke Scale (items 4 - 7)
3. Dietary history

Study procedures:

1. DEXA evaluation. Specific measurements will be made for lumbar spine, hip and distal radius; lateral vertebral assessment will be obtained if possible.

Biological Samples:

1. Two 10ml tubes of blood will be obtained from each participant. Serum will be separated and frozen in two aliquots to be saved for possible measurement of vitamin D levels (25OH vitamin D) and/or bone markers.

ELIGIBILITY:
Inclusion Criteria:

* History of brain injury at some defined time in the past (include stroke, traumatic brain injury, anoxia)
* Age 16 years and older (no upper age limit)
* Male and females
* Able to undergo a DEXA examination (able to lie on the DEXA table for 20-30 minutes)
* Able to provide answers to the questionnaires regarding medical and dietary history and demographics
* Able to provide informed consent

Exclusion Criteria:

* History of spinal cord injury
* History of traumatic brain damage
* Inability to lie down appropriately to obtain DEXA measurements
* Inability to communicate
* Anything condition that in the judgment of the physician would prevent the person from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have experienced brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern Univesity & Rehabilitation Institute of Chicago; Richard Harvey, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab; Elliot Roth, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Rehabilitation Institute of Chicago, Chicago, Illinois